CLINICAL TRIAL: NCT05419674
Title: Ten-day Amoxicillin-containing Dual Therapy as First-line Helicobacter Pylori Treatment in Elderly Patients: a Randomized Trial
Brief Title: Efficacy and Safety of Dual Therapy as First-line Treatment for Hp Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0323
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: dual therapy; bismuth-containing quadruple therapy; Helicobacter Pylori
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Rabeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- groupA: dual therapy (vonoprazan+amoxicillin) (Experimental): vonoprazan 20mg bid and amoxicillin 1000mg tid for 10 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- group B: dual therapy (rabeprazole+amoxicillin) (Experimental): rabeprazole 10mg tid and amoxicillin 1000mg tid for 10 days
  Interventions: Drug: Rabeprazole; Drug: Amoxicillin
- group C: bismuth-containing quadruple therapy (Active Comparator): rabeprazole 10 mg bid, colloidal bismuth pectin 200mg bid, amoxicillin 1000mg bid and clarithromycin 500mg bid for 10 days
  Interventions: Drug: Rabeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Colloidal bismuth pectin

INTERVENTIONS:
Drug: Vonoprazan — Potassium-competitive acid blocker
  Arms: groupA: dual therapy (vonoprazan+amoxicillin)
Drug: Rabeprazole — Proton pump inhibitor
  Arms: group B: dual therapy (rabeprazole+amoxicillin); group C: bismuth-containing quadruple therapy
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: Clarithromycin — Antibiotic for H. pylori eradication
  Arms: group C: bismuth-containing quadruple therapy
Drug: Colloidal bismuth pectin — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: group C: bismuth-containing quadruple therapy

SUMMARY:
This study aims to evaluate the efficacy of dual therapy compared with bismuth-containing quadruple therapy as first-line treatment for Helicobacter Pylori eradication, as well as the safety and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

1. having H. pylori related chronic gastritis confirmed by ¹³C-urea breath test, ¹⁴C-urea breath test and/or biopsy；
2. underwent gastroscopy within 1 year before treatment, liver and renal function tests and electrocardiogram within 3 months before treatment；
3. with no historical treatment for helicobacter pylori infection.

Exclusion Criteria:

1. administration of antibiotics, bismuth in 4 weeks prior to inclusion or antacids including H2 receptor antagonist, proton pump inhibitor and potassium-competitive acid blocker in 2 weeks prior to inclusion
2. with previous esophageal or gastric surgery
3. with severe systemic diseases, major organ like heart, lung, brain diseases, liver or kidney insufficiency, malignant tumor or other diseases
4. allergy to any of the study drugs
5. participated in other research within 3 months，cannot express his/her own ideas correctly or cannot cooperate with the researcher

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication Rate | Six to eight weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test six to eight weeks after completion of the medication. The eradication rates will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
Rate of Adverse Drug Reaction(ADR) | Within 7 days after completion of therapy
  Adverse drug reactions are classified into six types (with mnemonics): dose-related (Augmented), non-dose-related (Bizarre), dose-related and time-related (Chronic), time-related (Delayed), withdrawal (End of use), and failure of therapy (Failure).
Compliance Rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China